CLINICAL TRIAL: NCT02191618
Title: The WEB® Intrasaccular Therapy Study (WEB-IT)
Brief Title: The WEB-IT Clinical Study
Acronym: WEB-IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Microvention-Terumo, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP13-001
Record Dates: First submitted 2014-07-14; First posted 2014-07-16 (Estimated); Results first posted 2020-04-14 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2020-04

CONDITIONS: Wide Neck Bifurcation Intracranial Aneurysms; Intracranial Aneurysms
Keywords: Aneurysm; Intracranial Aneurysm; Vascular Diseases; Cardiovascular Diseases; Intracranial Arterial Diseases; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm; Vascular Diseases; Cardiovascular Diseases; Intracranial Arterial Diseases; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- WEB Aneurysm Embolization Device (Other): The WEB is an intra-aneurysmal device intended for use in endovascular embolization of intracranial aneurysms.
  The intended therapeutic effect of the WEB device is to line the neck of the aneurysm with a metallic structure that disrupts the inflow of blood, causing hemostasis within the aneurysm sac, and leading to thrombus formation within the implant.
  Interventions: Device: WEB

INTERVENTIONS:
Device: WEB — The WEB is an intra-aneurysmal device intended for use in endovascular embolization of intracranial aneurysms.
  Other Names: WEB Aneurysm Embolization Device

SUMMARY:
The study is a prospective, multicenter single-arm cohort. Patients with wide neck bifurcation aneurysms (WNBAs) have few choices for safe and effective endovascular treatment. In this study, all patients with qualifying WNBAs will be treated with the WEB. The primary effectiveness outcome of the study is the likelihood of complete intracranial aneurysm occlusion on the 1 year angiogram as adjudicated by a core laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥18 and ≤75 years.
* Patient must have a single ruptured or unruptured IA (intracranial aneurysm) requiring treatment.
* Patient must sign and date an IRB/EC-approved written informed consent prior to initiation of any study procedures.

Exclusion Criteria:

* Patient has an IA with characteristics unsuitable for endovascular treatment
* Patient has stroke-in-evolution within the prior 60 days
* Patient has had an SAH (subarachnoid hemorrhage) from a nonindex IA or any other intracranial hemorrhage within 90 days
* Patient's index IA was previously treated
* Patient is pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2023-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Arthur, MD, Principal Investigator — Methodist University Hospital, Memphis, TN; David Fiorella, MD, Principal Investigator — Stony Brook University, Stony Brook, NY
Locations (32):
- United States (26):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Sequent Medical, Aliso Viejo, California
  - Radiology Imaging Associates P.C., Englewood, Colorado
  - Lyerly Baptist, Inc, Jacksonville, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Louisville, Louisville, Kentucky
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Albany Medical Center, Albany, New York
  - Buffalo General Medical Center, Buffalo, New York
  - The Mount Sinai Medical Center, New York, New York
  - Stony Brook University, Stony Brook, New York
  - Carolina NeuroSurgery & Spine Associates, P.A., Charlotte, North Carolina
  - Riverside Methodist Hospital/ Ohio Health Research Institute, Columbus, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Ft. Sanders Regional Medical Center, Knoxville, Tennessee
  - Methodist University Hospital, Memphis, Tennessee
  - Baptist Memorial Hospital, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah Medical Center, Salt Lake City, Utah
  - West Virginia University, Morgantown, West Virginia
- Royal University Hospital, Saskatoon, Saskatchewan, Canada
- Rigshospitalet, Copenhagen, Denmark
- Helios Hospital, Erfurt, Germany
- National Institute of Neurosciences, Budapest, Hungary
- Turkey (Türkiye) (2):
  - Koru Hospital, Ankara
  - Marmara University Faculty of Medicine Pendik Training and Research Hospital, Istanbul

REFERENCES:
- [Derived] Arthur AS, Molyneux A, Coon AL, Saatci I, Szikora I, Baltacioglu F, Sultan A, Hoit D, Delgado Almandoz JE, Elijovich L, Cekirge S, Byrne JV, Fiorella D; WEB-IT Study investigators. The safety and effectiveness of the Woven EndoBridge (WEB) system for the treatment of wide-necked bifurcation aneurysms: final 12-month results of the pivotal WEB Intrasaccular Therapy (WEB-IT) Study. J Neurointerv Surg. 2019 Sep;11(9):924-930. doi: 10.1136/neurintsurg-2019-014815. Epub 2019 Apr 16. PMID 30992395
- [Derived] Fiorella D, Molyneux A, Coon A, Szikora I, Saatci I, Baltacioglu F, Sultan A, Arthur A; WEB-IT Study Investigators. Demographic, procedural and 30-day safety results from the WEB Intra-saccular Therapy Study (WEB-IT). J Neurointerv Surg. 2017 Dec;9(12):1191-1196. doi: 10.1136/neurintsurg-2016-012841. Epub 2017 Jan 17. PMID 28096478

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | WEB Aneurysm Embolization Device
Started | 150
Completed | 143
Not Completed | 7
Not completed — Withdrawal by Subject | 3
Not completed — Missed Visit | 4

BASELINE CHARACTERISTICS:
Arm/Group | WEB Aneurysm Embolization Device
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.98 (10.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 40
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not obtained for subjects from the European and Canadian sites.
  Participants
    American Indian or Alaska Native | 0
    Asian | 4
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 14
    White | 98
    More than one race | 0
    Unknown or Not Reported | 34
Region of Enrollment [Number; unit: participants]
  United States | 116
  Turkey | 20
  Hungary | 10
  Canada | 2
  Denmark | 1
  Germany | 1

OUTCOME MEASURES:

1. Primary Outcome: The Primary Safety Endpoint Included Any Death or Major Stroke in the First 30 Days and Neurologic Death or Ipsilateral Major Stroke Between Day 31 and Day 365.
Description: The study's primary safety endpoint was the proportion of subjects with death of any nonaccidental cause or any major stroke (defined as an ischemic or hemorrhagic stroke resulting in an increase of 4 points or more on the National Institutes of Health Stroke Scale (NIHSS)) within the first 30 days after treatment or major ipsilateral stroke or death due to neurologic cause from day 31 to 365 days after treatment.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | WEB Aneurysm Embolization Device
Number analyzed (Participants) | 150
Participants | 1

2. Primary Outcome: Percentage of Subjects With Complete Aneurysm Occlusion Assessed Using the WEB Occlusion Scale (WOS) Without Retreatment, Recurrent Subarachnoid Hemorrhage, Without Significant Parent Artery Stenosis (>50% Stenosis) at One Year After Treatment
Description: The primary effectiveness endpoint was defined as the percentage of subjects with complete aneurysm occlusion assessed using the WEB Occlusion Scale (WOS) without retreatment, recurrent subarachnoid hemorrhage, without significant parent artery stenosis (>50% stenosis) at one year after treatment in the mITT population.
Time Frame: 12 months
Population: The overall number of participants analyzed is 143 due to 3 subjects withdrawing and 4 subjects that missed their 1 year follow up visit.
Measure: Count of Participants; unit: Participants
Arm/Group | WEB Aneurysm Embolization Device
Number analyzed (Participants) | 143
Participants | 77

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- CEC Adjudicated Adverse Events Through 1-Year: The WEB is an intra-aneurysmal device intended for use in endovascular embolization of intracranial aneurysms.
  The intended therapeutic effect of the WEB device is to line the neck of the aneurysm with a metallic structure that disrupts the inflow of blood, causing hemostasis within the aneurysm sac, and leading to thrombus formation within the implant.
Arm/Group | CEC Adjudicated Adverse Events Through 1-Year
All-Cause Mortality (participants affected / at risk) | 0/150
Serious Adverse Events (participants affected / at risk) | 33/150
Other Adverse Events (participants affected / at risk) | 54/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CEC Adjudicated Adverse Events Through 1-Year (N=150)
Angina pectoris (Cardiac disorders) | 1 (4)
Cardiac arrest (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2)
Cushing's syndrome (Endocrine disorders) | 1 (2)
Crohn's disease (Gastrointestinal disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Benign intracranial hypertension (Nervous system disorders) | 1 (1)
Confusional state (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Ischemic Stroke (Nervous system disorders) | 6 (7)
Seizure (Nervous system disorders) | 2 (2)
Subarachnoid hemorrhage (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
TIA (Nervous system disorders) | 3 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vessel puncture site hematoma (Surgical and medical procedures) | 4 (4)
Arterial thrombosis (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (3)
Vascular occlusion (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CEC Adjudicated Adverse Events Through 1-Year (N=150)
Nausea (Gastrointestinal disorders) | 10 (11)
Vessel puncture site hematoma (Vascular disorders) | 8 (8)
Headache (Nervous system disorders) | 36 (44)
Adverse drug reaction (General disorders) | 14 (15)
Visual impairment (Eye disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-08-12): https://cdn.clinicaltrials.gov/large-docs/18/NCT02191618/Prot_000.pdf
  • Statistical Analysis Plan (2015-08-12): https://cdn.clinicaltrials.gov/large-docs/18/NCT02191618/SAP_001.pdf